CLINICAL TRIAL: NCT05895578
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of a Probiotic on the Urinary Tract Microbiota in Women With Recurrent Urinary Tract Infections (rUTI).
Brief Title: Effect of a Probiotic on the Urinary Tract Microbiota of Participants With Recurrent Urinary Tract Infection.
Acronym: PROBUTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTI/23.01
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Probiotic (Active Comparator): 2 Capsule daily containing approximately 1*10E9 colony forming unit (CFU) of Lactobacillus CECT 9422 +1*10E9 colony forming unit (CFU) of Bifidobacterium CECT 30257.
  Interventions: Dietary Supplement: Probiotic
- Probiotic + placebo (Active Comparator): One capsule daily containing approximately 1*10E9 colony forming unit (CFU) of Lactobacillus CECT 9422 +1*10E9 colony forming unit (CFU) of Bifidobacterium CECT 30257 and 1 capsule of placebo supplement.
  Interventions: Dietary Supplement: Probiotic + placebo
- Placebo (Placebo Comparator): Two capsules daily of Placebo supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 1 capsule of probiotic (Lactobacillus CECT 9422 + Bifidobacterium CECT 30257) every 12 hours for 6-months.
  Arms: Probiotic
Dietary Supplement: Probiotic + placebo — 1 capsule of probiotic + 1 capsule of placebo per day for 6-months.
  Arms: Probiotic + placebo
Dietary Supplement: Placebo — 1 capsule of placebo every 12 hours for 6-months.
  Arms: Placebo

SUMMARY:
Urinary tract infections (UTIs) are the most common bacterial infections in women. 50% of women experiencing at least one UTI in their lifetime with an annual prevalence of 0.5-0.7%.

An interventional, randomized, double-blind, placebo-controlled study will be conducted to investigate the effect of a probiotic strains on the urinary tract microbiota in participants with recurrent urinary tract infection (rUTI).

The study duration will be 6 and a half months, including 6 months product intake. Participants will be randomly assigned to one of the three study groups: control group with placebo administration, probiotic administration group (1 dose) and probiotic administration group (2 doses).

ELIGIBILITY:
Inclusion Criteria:

* Adult women with aged between 18 and 55 years old, diagnosed with recurrent UTI (defined as at least two episodes during the last six months or three during the last 12 months).
* Diagnosed, the last 7days, for a new UTI episode.
* Written informed consent signed.

Exclusion Criteria:

* Menopausal
* Pregnant, breastfeeding or planning to become pregnant during the study.
* Congenital abnormalities of the urinary tract.
* Renal functional alterations, such as neurogenic bladder or vesicoureteral reflux.
* Relevant renal disorders, such as interstitial cystitis, renal lithiasis, renal failure, kidney transplantation, pyelonephritis, renal nephropathy, etc.
* Permanent catheter.
* Immunocompromised (eg: cancer and/or transplant, patients who are taking immunosuppressive drugs, patients with hereditary diseases that affect or may affect the immune system).
* Type I diabetes.
* With a defect in the intestinal epithelium barrier (eg: chronic diarrhea, inflammatory bowel disease).
* Heart failure and cardiac medical history (eg, artificial heart valve, medical history of infective endocarditis, rheumatic fever, or cardiac malformation).
* Under antibiotics prophylactic treatment without willingness to leave it at the time of inclusion.
* Probiotics supplementation during the previous 2 weeks.
* To have received Urovac, Uro-Vaxom or equivalent vaccine during the last year.
* Currently participating in another clinical trial.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the number of participants with a positive urine culture | Before intervention
  The number of participants with a positive urine culture will be compared between groups of treatment.
Evaluate the number of participants with a positive urine culture | After 3 months of intervention.
  The number of participants with a positive urine culture will be compared between groups of treatment.
Evaluate the number of participants with a positive urine culture | After 6 months of intervention.
  The number of participants with a positive urine culture will be compared between groups of treatment.
Evaluate the total bacterial count in urine samples. | Before intervention
  The total bacterial count in urine samples will be compared between groups of treatment.
Evaluate the total bacterial count in urine samples. | After 3 months of intervention
  The total bacterial count in urine samples will be compared between groups of treatment.
Evaluate the total bacterial count in urine samples. | After 6 months of intervention
  The total bacterial count in urine samples will be compared between groups of treatment.

SECONDARY OUTCOMES:
Number of UTI episodes | After 3 and 6 months of intervention.
Infection free participants (%) | After 6 months of intervention.
Elapsed time until the 1st episode of UTI. | After 6 months of intervention.
Elapsed time between the 1st and 2nd episode of UTI. | After 6 months of intervention.
Elapsed time between the 2nd and 3rd episode of UTI. | After 6 months of intervention.
Duration of UTI episodes. | After 6 months of intervention.
The number of participants which associate sexual activity with the UTI episodes | After 6 months of intervention.
  The number of participants which associate sexual activity with the apperance of an UTI episode will be counted and compared between groups.
Number of present symptoms during new UTI episodes. | After 6 months of intervention.
Number of participants with dysuria. | After 6 months of intervention.
Duration of dysuria. | After 6 months of intervention.
Number of participants with pollakiuria | After 6 months of intervention.
Duration of pollakiuria | After 6 months of intervention.
Number of participants with urinary urgency. | After 6 months of intervention.
Duration of urinary urgency. | After 6 months of intervention.
Number of participants with tenesmus. | After 6 months of intervention.
Duration of tenesmus. | After 6 months of intervention.
Number of participants with hematuria. | After 6 months of intervention.
Duration of hematuria | After 6 months of intervention.
Number of participants with dyspareunia | After 6 months of intervention.
Duration of dyspareunia | After 6 months of intervention.
Number of participants with pelvic pain | After 6 months of intervention.
Duration of pelvic pain | After 6 months of intervention.
Number of participants with fever (Tª ≥ 38ºC). | After 6 months of intervention.
Duration of fever (Tª ≥ 38ºC). | After 6 months of intervention.
Number of participants with cloudy and smelly urine | After 6 months of intervention.
Duration of cloudy and smelly urine | After 6 months of intervention.
Number of antibiotics administered for the UTI episode. | After 6 months of intervention.
Duration of antibiotic treatment for the UTI episode. | After 6 months of intervention.
Number of antibiotic treatments administered during new UTI episodes. | After 6 months of intervention.
Duration of antibiotic treatments administered during new UTI episodes. | After 6 months of intervention.
Microbiome composition of stool samples determined by 16S sequencing. | After 6 months of intervention.
  The composition of fecal microbiome will be compared between treatments group and time
Microbiota composition of urine samples determined by culture techniques. | After 6 months of intervention.
  The composition of urine microbiota will be compared between treatments group and time.
Metabolomic profile of urine samples. | After 6 months of intervention.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital La Moraleja, Madrid
  - Hospital La Zarzuela, Madrid
  - Hospital San Francisco de Asís, Madrid